Study Title: Best Practice With Rocuronium, Neostigmine, Sugammadex, and Subjective Monitoring

NCT03543826

Document title: Statistical Analysis Plan

Date of the document: 5/8/2019

## Statistical analysis

We present descriptive statistics [mean (standard deviation) or frequencies] for baseline measures of patient and surgery characteristics. The primary endpoint, incidence of PRNB (nTOFR <0.9) on arrival to the PACU, was calculated with exact binomial 95% confidence interval, and graphically displayed using scatterplots. The primary analysis was "per-protocol" and patients were excluded if the protocol was not followed. Secondary endpoints included severe PRNB, defined as nTOFR <0.7 on arrival to the PACU, and PRNB at time of tracheal extubation (nTOFR <0.9). These were also calculated with the exact confidence intervals. Additionally, we calculated the incidence of severe PRNB at time of tracheal extubation and the incidence of PRNB using raw (non-normalized) measurements.

We compared the duration between end of surgery and arrival to the PACU for patients whose tracheas were extubated in the OR and those extubated in PACU. We also compared the duration between end of surgery and arrival to the PACU for patients receiving sugammadex or neostigmine.